CLINICAL TRIAL: NCT03257969
Title: Impact of the DROP (Drug Related Problems in Oncology Practice) Program of Pharmaceutical Interventions of the French Society of Oncological Pharmacology Versus Usual Care on the DRP (Drug Related Problems) Related to Oral Anticancer Drugs in Ambulatory Patients with Risk Factors
Brief Title: Impact of the DROP Program on the DRP (Drug Related Problems) Related to Oral Anticancer Drugs in Ambulatory Patients with Risk Factors
Acronym: DROP-SFPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL17_0029
Record Dates: First submitted 2017-07-27; First posted 2017-08-22 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Cancer
Keywords: Oral chemotherapy; Health related program; Secured drug intake; Pharmacist intervention; Cancer outpatient
MeSH Terms: conditions — Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The DROP program (Experimental)
  Interventions: Behavioral: The DROP program of pharmaceutical interventions
- Standard of care (Other)
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: The DROP program of pharmaceutical interventions — Multidisciplinary program that includes informative sessions with a hospital pharmacist about the oral anticancer drug: information is given to the patient on adverse events occurrence and there management; and optimizing drug dosage plan, including drug-drug interactions.
  Arms: The DROP program
Behavioral: Standard of care — In the group with standard of care, patients will have interviews with a clinical research associate only dedicated to the record of data for outcomes assessment.
  Arms: Standard of care

SUMMARY:
The rise of oral anticancer drugs favors outpatient care but exposes patients to new risks compared to injectable chemotherapy at hospital: non-adherence to treatment, inappropriate management of side effects and interactions with other co-prescribed drugs. Latrogenic risk of these treatments is reinforced in older patients with frequent comorbidities, taking multiple pharmaceutical treatments for long periods and followed by several prescribers.

The literature reports an emergence of drug related problems (DRP) in more than 90% of patients, with an average number of 0 to 4 per patient. The clinical consequences (reduced efficacy and potentiation of toxicity) are all the more important that outpatient monitoring of treatments prescribed at the hospital remains underdeveloped due to default of coordination between these two settings.

Medical care and prevention of these DRP are difficult because of a lack of information and tools shared between hospital and liberal actors. Experiments are developed according to different organizational models, frequently focused on the pharmaceutical analysis of prescriptions, the detection of DRP and their control, but they stay still undervalued. In this context, the French Society of Oncological Pharmacology (SFPO - Société Française de Pharmacie Oncologique) provides to hospital and ambulatory care pharmacists the Oncolien website and proposes to assess the impact of a program of pharmaceutical interventions named DROP. The hypothesis of the study is that the DROP program will secure the medical care of patients with oral anticancer drugs compared to the usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years old or more
* With cancer
* For wich the initiation or change of an oral anticancer drug is prescribed
* With life expectancy estimated to be 6 months or more, in the opinion of the investigator
* Of which the treatment with oral anticancer medication is estimated to be 6 months or more in the opinion of the oncologist
* Benefiting from an initiation or a change of oral anticancer agents according to the MA: cytotoxic agent, targeted therapy, hormonal therapy (excluding adjuvant treatments);
* of which the oral anticancer drug is delivered in pharmacy of town or in retrocession hospital;
* With ambulatory status (not hospitalized for the management and treatment )
* Taking 5 or more drugs, including the oral anticancer treatment, and / or treated with an oral anticancer drug requiring complex regimen (combination of 2 oral anticancer drugs, or sequential rate of intake, or associated to intravenous chemotherapy)
* With a sufficient autonomy for the management of medication at home
* Without either cognitive disorders or major psychiatric disorders, in the opinion of the investigator
* Ability to read, write and understand the French language
* Having given his written consent to participate in the study
* Patient affiliated to the social security scheme or equivalent

Exclusion Criteria:

* Pregnant or lactating woman
* Patient on anti-PD1, anti-PDL-1 or anti-CTLA4-4 immunotherapy concomitant with oral anticancer treatment
* Patient under radiotherapy concomitant treatment with oral anticancer
* Oral anticancer agent prescribed in a delivery circuit as part of an ATU or clinical trial;
* Patient with significant cognitive or psychiatric disorders, in the opinion of the investigator;
* Management of drug treatment at home is performed exclusively by the caregiver;
* Not having declared a doctor;
* Not having a usual city pharmacy, or reporting 2 or more usual city pharmacies;
* Patient who has already benefited from a therapeutic education program
* In institution or guardianship, major protected by the Law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2019-06-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of DRP (Drug Relates Problems) related to oral anticancer drugs per patient, in total and for each category | 9 months post-inclusion
  DRP are defined as the number of: adverse reactions (grade 2-3-4); drug interactions (contraindication, association not recommended, precautionary use); and medication errors with proven harm or requiring appropriate monitoring (Medication Error Index of the National Coordinating Council for Medication Error Reporting and Prevention, grade D to I).

SECONDARY OUTCOMES:
Total number of DRP related to all prescribed drugs per patient | 6 months and 9 months post-inclusion
  DRP are defined as the number of: adverse reactions (grade 2-3-4); drug interactions (contraindication, association not recommended, precautionary use); and medication errors with proven harm or requiring appropriate monitoring (Medication Error Index of the National Coordinating Council for Medication Error Reporting and Prevention, grade D to I).
Number of adaptations in the prescription of oral anticancer drugs, related to DRP, per patient | 6 months and 9 months post-inclusion
  dose adjustments, cure spacing, interruptions and cessation of treatment.
Relative dose intensity of the oral anticancer drug | 6 months post-inclusion
  Relative dose intensity will be computed by the ratio between the overall dose prescribed during the 6 months of follow-up and the theoretical dosage according to the summary of product characteristics of the market authorization.
Adherence to the oral anticancer drug | 6 months post-inclusion
  Adherence will be measured with the Girerd questionnaire score 6 items from the Ameli Health Insurance website and the rate of prescription renewal by the ambulatory pharmacy (adherence will be defined as a rate ≥80%).
Number of imaging acts and nature of acts | During the 6 months of follow-up
  To evaluate consumption of unscheduled ambulatory care related to DRP
Number of acts of biology and nature of acts | During the 6 months of follow-up
  To evaluate consumption of unscheduled ambulatory care related to DRP
Number of medical consultations | During the 6 months of follow-up
  To evaluate consumption of unscheduled ambulatory care related to DRP
Number of prescriptions of drugs (without prescription of the oral anticancer drug) and nature of these drugs | During the 6 months of follow-up
  To evaluate consumption of unscheduled ambulatory care related to DRP
Number of hospital admissions | During the 6 months of follow-up
  To evaluate unplanned hospital admissions related to DRP
Patient's quality of life, measured with the EuroQol 5-Dimensions questionnaire | At inclusion and 6 months from the treatment initiation
Patient's satisfaction with treatment, measured with the SAT-MED Q questionnaire | At inclusion and 6 months from the treatment initiation
Health locus of control, measured with the Therapeutic Self Care Toll (TSCT) scale | At inclusion and 6 months from the treatment initiation
Number of interventions of primary care actors with the patient | During the 9 months of follow-up
  To evaluate the involvement of primary care actors in the DROP program
Number of time the Oncolien website was used by ambulatory care pharmacists | During the 9 months of follow-up
  To evaluate the involvement of primary care actors in the DROP program
Number of forms helping the delivery of the oral anticancer drug used by ambulatory care pharmacists | During the 9 months of follow-up
  To evaluate the involvement of primary care actors in the DROP program
Number of patient-advice forms downloaded and delivered to the patient | During the 9 months of follow-up
  To evaluate the involvement of primary care actors in the DROP program
Number and reason for solicitations of hospital actors by the primary care actors, in the context of information sharing | During the 9 months of follow-up
  To evaluate the involvement of primary care actors in the DROP program
Patient's satisfaction for the DROP program | At 9 months post-inclusion
  Satisfaction will be measured with a 10-point visual analog scale.
Ambulatory care physician's and pharmacist's satisfactions with the DROP program | At 9 months post-inclusion
  Satisfaction will be measured with a 10-point visual analog scale.
Efficiency of the DROP program | 9 months post-inclusion
  Efficiency will be computed by the incremental cost-efficacy ratio between the DROP program and the usual care.

CONTACTS AND LOCATIONS:
Locations (1):
- Service pharmaceutique, Unité de Pharmacie Clinique Oncologique, Centre Hospitalier Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ranchon F, Huot L, Bardin C, Madelaine I, Cazin JL, Pourroy B, Tilleul P, Lemare F, Rioufol C. Randomised controlled trial to assess the impact of hospital-community pharmaceutical care on drug-related problems in oncology practice for at-risk outpatients treated with oral anticancer drugs-a French Society for Oncology Pharmacy (SFPO) study: DROP-SFPO study protocol. BMJ Open. 2025 Jun 27;15(6):e094825. doi: 10.1136/bmjopen-2024-094825. PMID 40578885